CLINICAL TRIAL: NCT01262807
Title: Reducing Range of Motion Deficits With In-cast Exercises: A Randomized Controlled Trial
Brief Title: Reducing Range of Motion Deficits Post Radial Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Pan Am Clinic (Other)
Responsible Party: Jamie Dubberley, University of Manitoba
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: H2010:187
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Radius Fractures
Keywords: fracture; radius; adult; range of motion
MeSH Terms: conditions — Radius Fractures; Fractures, Bone | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): This group will receive instructions on specific exercises to perform after randomization.
  Interventions: Other: Exercises
- Standard Care (No Intervention): This group will receive standard care

INTERVENTIONS:
Other: Exercises — A specific set of standardized exercises will be taught to patients who are randomized to the intervention group. They will be instructed to do these exercises daily while in-cast. They will have an exercise log to track adherence.
  Arms: Exercise

SUMMARY:
This a randomized controlled study to test the hypothesis that patients who perform in-cast exercises will have superior range of motion immediately post-cast removal, without a concomitant increase in complication rate when compared with a control group who receives standard post cast care which does not include the intervention exercises.

ELIGIBILITY:
Inclusion Criteria:

* patient experienced distal radial fracture
* patient is over 18 years of age
* patient can follow instructions and comply with protocol
* fracture is managed non-operatively

Exclusion Criteria:

* bilateral wrist fractures
* previous fracture to the affected wrist
* previous range of motion limitations to the affected wrist
* involvement of other upper extremity structures (i.e. shoulder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in range of motion | 6 weeks, 6 months, 1 year

SECONDARY OUTCOMES:
Complications | 6 weeks
  The number and type of complications will be collected and compared between groups

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Dubberley, MD, Principal Investigator — University of Manitoba; Jeff Leiter, PhD, Study Chair — Pan Am Clinic; Kristy Wittmeier, PhD, Study Director — Winnipeg Health Sciences Centre
Locations (1):
- Pan Am Clinic, Winnipeg, Manitoba, Canada